CLINICAL TRIAL: NCT01763944
Title: A Randomized Controlled Clinical Trial of Carbohydrate Restriction Among Men With A Rising PSA After Failed Primary Therapy for Prostate Cancer
Brief Title: Carbohydrate Restriction and Prostate Cancer Growth
Acronym: CAPS2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH); Robert C. Atkins Foundation (Other); Cedars-Sinai Medical Center (Other); Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00041857; 1K24CA160653-01A1 (NIH); 192822 (Other Grant/Funding Number: Atkins Foundation)
Record Dates: First submitted 2012-12-14; First posted 2013-01-09 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: diet; prostate cancer; carbohydrate; lifestyle
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Diet, Carbohydrate-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low carbohydrate, lifestyle counseling (Active Comparator): The Low carbohydrate arm will receive counseling to follow a carbohydrate restriction diet (<20 grams per day) for 6 months.
  Interventions: Behavioral: Low carbohydrate diet
- Control (No Intervention): The control arm will receive no dietary intervention.

INTERVENTIONS:
Behavioral: Low carbohydrate diet — The Low carbohydrate diet intervention recommends patients to limit carbohydrate intake to less than 20 gram per day.
  Arms: Low carbohydrate, lifestyle counseling

SUMMARY:
No treatments have been shown to slow prostate cancer progression after radical prostatectomy. We hypothesize that a carbohydrate restricted diet will slow prostate cancer growth. A total of 60 men with a rising prostate-specific antigen (PSA) after failed primary treatment will be recruited and randomized to either a low-carbohydrate diet (<20 grams carbohydrates/day) or a no-diet control (standard of care) for 6 months. The primary outcome is PSA doubling time.

ELIGIBILITY:
Inclusion Criteria:

* Received prior radical prostatectomy or definitive local radiation for prostate cancer (either external beam radiation, brachytherapy, or combination)
* PSA within the past 3 months is between 0.4 and 20 if prior radical prostatectomy, or between 3 and 20 ng/ml if prior radiation therapy.
* PSA doubling time (PSADT) >3 months and <36 months

  1. Calculated based at least 2 values (at least 0.2) in the prior 2 years with the first and last PSA separated by at least 3 months
  2. Use all values in the last 2 years to calculate PSADT
  3. PSADT calculated while NOT on androgen deprivation therapy (ADT).
  4. If prior ADT use, then documented either A) normal testosterone or B) a testosterone within 50 points of normal and stable (defined as a second testosterone at least 6 weeks later that is equal or lower than the first testosterone) is required before starting to calculate PSADT.
* BMI >=24 kg/m2
* Willing to be randomized to a no-diet control or a low-carbohydrate diet
* Reads, writes, and understands English

Exclusion Criteria:

* Anticipate needing secondary prostate cancer therapy within the next 6 months (i.e. radiation, or hormonal therapy)
* Current use of weight loss medications including herbal weight loss supplements or enrolled in a diet/weight loss program
* Currently on therapy aimed at lowering testosterone levels (includes gonadotropin-releasing hormone (GnRH) agonist/antagonist, prior bilateral orchiectomy, oral anti-androgens, or 5-alpha reductase inhibitors). Testosterone replacement is allowed but treatment should be stable during the entire study.
* Known distant metastatic disease
* Already consuming a carbohydrate-restricted or vegetarian diet
* Unable or unwilling to adhere to a carbohydrate-restricted dietary intervention
* Weight loss >5% of body weight in the last 6 months
* Medical comorbidities that in the opinion of the investigator limits the patient's ability to complete this study

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-20 (Actual)

PRIMARY OUTCOMES:
PSA doubling time (change in PSA over time) | Baseline, 3 and 6 months
  PSA doubling time will be estimated from PSA measured at baseline, 3 and 6 months post randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Pao-Hwa Lin, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Duke University Medical Center, Durham, North Carolina
  - Durham VA Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Lin PH, Howard L, Freedland SJ. Weight loss via a low-carbohydrate diet improved the intestinal permeability marker, zonulin, in prostate cancer patients. Ann Med. 2022 Dec;54(1):1221-1225. doi: 10.1080/07853890.2022.2069853. PMID 35486445
- [Derived] Lin PH, Howard L, Freedland SJ. Impact of Low Carbohydrate Diet on Self-Report Fatigue and Weakness in Prostate Cancer Patients. J Urol. 2021 Sep;206(3):499-501. doi: 10.1097/JU.0000000000001780. Epub 2021 Apr 5. No abstract available. PMID 33819069
- [Derived] Freedland SJ, Allen J, Jarman A, Oyekunle T, Armstrong AJ, Moul JW, Sandler HM, Posadas E, Levin D, Wiggins E, Howard LE, Wu Y, Lin PH. A Randomized Controlled Trial of a 6-Month Low-Carbohydrate Intervention on Disease Progression in Men with Recurrent Prostate Cancer: Carbohydrate and Prostate Study 2 (CAPS2). Clin Cancer Res. 2020 Jun 15;26(12):3035-3043. doi: 10.1158/1078-0432.CCR-19-3873. Epub 2020 Feb 27. PMID 32108029